CLINICAL TRIAL: NCT01447589
Title: A Phase I Dose Escalation Study of the HIV Protease Inhibitor, Nelfinavir, Given Concomitantly With Radical Radiotherapy (RT) for the Treatment of Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Radical Lung Radiotherapy Plus Nelfinavir
Acronym: NelfLung
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: failed to recruit, no suitable patients
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Linda Ward, QA Coordinator, Cancer Centre, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP-TSC-651
Record Dates: First submitted 2011-07-18; First posted 2011-10-06 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: Radiosensitiser
MeSH Terms: conditions — Lung Neoplasms | interventions — Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nelfinavir plus radical radiotherapy (Experimental): Nelfinavir given in combination with radical RT
  Interventions: Drug: nelfinavir; Radiation: Radical Radiotherapy

INTERVENTIONS:
Drug: nelfinavir — Nelfinavir tablets BD 7 days per week from D-7 of starting radiotherapy until completion of radiotherapy on D47. 3 dose levels: 750 mg bd; 1000 mg bd; and 1250 mg bd.
  Other Names: Viracept®
Radiation: Radical Radiotherapy — Total dose of 66 Gy delivered in 33 fractions (2.0 Gy/fraction) to the primary tumour plus a margin.

SUMMARY:
The aim of this clinical trial is to test whether the drug nelfinavir, which can increase the effectiveness of radiotherapy, can be given safely at the same time as a full dose of radiotherapy for lung cancer.

It is thought that one way that nelfinavir works is through causing changes in the blood vessels within tumours. The status of tumour blood vessels and the blood flow through them will be investigated during the trial using special imaging techniques. The dose of radiation used in this trial is greater than that used in previous trials with nelfinavir in other disease settings and the response of normal lung to the combination of nelfinavir plus radiation is unknown. Therefore, a low dose of nelfinavir will be given to the first few patients that participate and will be gradually increased in subsequent groups of patients provided that no worrying side effects are identified. There is a single report of serious side-effects in an AIDs patient who was treated with radiotherapy for lung cancer when he was also taking nelfinavir. However, in this case nelfinavir was taken at a dose 3-fold higher than the highest dose level to be tested in this trial. An important goal of this trial is to select the optimum dose of nelfinavir to be used in combination with lung radiotherapy, that can then be tested more extensively in future trials.

The radiotherapy treatment in this trial has been carefully designed to minimise the amount of healthy lung that receives radiation. Some specialised imaging techniques will be used during radiotherapy planning and delivery to help ensure that the lung cancer is targeted very precisely by radiation and that normal lung is avoided as much as possible.

One effect of nelfinavir is to interfere with the function of a particular protein in cells (called AKT). The degree to which this happens can be measured in cells from blood or tissue samples. Therefore, another aim of the study is to investigate AKT and related proteins, to check whether nelfinavir is having the predicted effect.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC except bronchoalveolar cancer
* Patients deemed suitable for radical RT according to local policy
* TNM stage T1-2, N0-1, M0 plus patients with local recurrence
* Adequate lung function as defined by protocol
* Age ≥ 18 years
* ECOG performance status 0-2
* Written informed consent
* Patient able and willing to comply with all protocol requirements

Exclusion Criteria:

* History of other active invasive malignancy (excluding non-melanoma skin cancer and in situ carcinoma of the cervix), where the extent of disease or treatment for that condition may interfere with the study endpoints
* Previous RT to the chest
* Chemotherapy, immunotherapies or investigational medicinal products within 4 weeks of the start of nelfinavir treatment. Ie any neoadjuvant treatment must be completed 4 weeks prior.
* Liver impairment (serum bilirubin ≥ 2 times upper limit of normal, serum AST ≥ 2 times the upper limit of normal)
* Pregnant or breast-feeding women or women of childbearing potential unless effective methods of contraception are used. Contraceptives that contain norethisterone or ethinylestradiol must be replaced by other contraceptive measures
* Concurrent use of contraindicated drugs that cannot be substituted or discontinued 2 weeks or more prior to the start of trial treatment
* Known hypersensitivity to nelfinavir or any of its excipients
* Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | One year
  To establish the maximum tolerated dose of nelfinavir in combination with radical radiotherapy for patients with non-small cell lung cancer

SECONDARY OUTCOMES:
Number of participants with adverse events | One year
  To assess the safety profile of combined nelfinavir together with radiotherapy in patients with NSCLC.
Radiotherapy control rate | 3 and 12 months
  To determine in-field radiotherapy treatment control rate at 3 and 12 months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Vallis, Principal Investigator — University of Oxford and Oxford Radcliffe NHS Trust
Locations (1):
- Oxford Radcliffe NHS Trust, Oxford, Oxfordshire, United Kingdom